CLINICAL TRIAL: NCT05910164
Title: Single-center, Randomized, Crossover Clinical Study to Assess Patient Preference Between the Use of a Prefilled Syringe or a Prefilled Pen Device for Pegfilgrastim Administration (PELGRAZ) as Primary Prophylaxis of Chemotherapy-related Neutropenia
Brief Title: Patient Preference Between a Prefilled Syringe or a Prefilled Pen Device for Administration of Pegfilgrastim
Acronym: PELGRAZ
Status: Completed | Type: Observational
Sponsor: Institut Rafael (Other)
Responsible Party: Sponsor
Other Study IDs: IR-2022/0011; ID RCB: 2022-A01465-38 (Other: ANSM France)
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-09

CONDITIONS: Patient Preference; Febrile Neutropenia, Drug-Induced; Patient Satisfaction
Keywords: patient preference; pegfilgrastim; chemotherapy prophylaxis; febrile neutropenia; survey; questionnaires
MeSH Terms: conditions — Patient Preference; Chemotherapy-Induced Febrile Neutropenia; Patient Satisfaction; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A) administration starting with prefilled syringe: - Group A = Phase 1 then phases 2, 3, 4
  The study protocol consists of 4 different stages
  * Phase 1: injection by pre-filled syringe by a state-certified nurse (IDE)
  * Phase 2: pen injection guided (thanks to the detailed information) by the IDE
  * Phase 3: injection by pen in autonomy supervised by the IDE (can only interfere in case of non-compliance with the injection protocol) = Learning phase
  * Phase 4: injection by pen in complete autonomy, patient alone
  Interventions: Device: PELGRAZ prefilled syringe or PELGRAZ prefilled pen
- B) administration starting with prefilled pen: - Group B = Phase 2, 3, 4 then phase 1
  The study protocol consists of 4 different stages
  * Phase 1: injection by pre-filled syringe by a state-certified nurse (IDE)
  * Phase 2: pen injection guided (thanks to the detailed information) by the IDE
  * Phase 3: injection by pen in autonomy supervised by the IDE (can only interfere in case of non-compliance with the injection protocol) = Learning phase
  * Phase 4: injection by pen in complete autonomy, patient alone
  Interventions: Device: PELGRAZ prefilled syringe or PELGRAZ prefilled pen

INTERVENTIONS:
Device: PELGRAZ prefilled syringe or PELGRAZ prefilled pen — PELGRAZ prefilled syringe or PELGRAZ prefilled pen https://www.ema.europa.eu/en/medicines/human/EPAR/pelgraz

SUMMARY:
Febrile neutropenia (NF) is a common serious complication of cancer chemotherapy. Outpatient management of chemotherapy treatments is made essential by the volume of patients treated, respect for their quality of life and the lack of hospitalization resources.

The prevention of NF is well documented and its success depends on the risks of developing NF related to the type of chemotherapy protocol used and the profile of the patient and his disease.

Pegfilgrastim (G-CSF, biosimilar medicine) injection has been shown to prevent (febrile) neutropenia. It is routinely prescribed on an outpatient basis for patients treated with chemotherapy (CT), several thousand times a year in our geographical area.

In order to take into account patient preferences and help clinical decision-making, this study will be conducted on the basis of self-administered questionnaires. The aim of the research is to assess patient preference for receiving administration of PELGRAZ (Accord Healthcare) using a prefilled syringe or a prefilled pen device. In a second step, this study will evaluate the learning of the patient and his autonomy during a pen self-injection guided by a nurse.

DETAILED DESCRIPTION:
Febrile neutropenia (NF) is a common serious complication of cancer chemotherapy. Outpatient management of chemotherapy treatments is made essential by the volume of patients treated, respect for their quality of life and the lack of hospitalization resources.

The prevention of NF is well documented and its success depends on the risks of developing NF related to the type of chemotherapy protocol used and the profile of the patient and his disease.

Pegfilgrastim (G-CSF, biosimilar medicine) injection has been shown to prevent (febrile) neutropenia. It is routinely prescribed on an outpatient basis for patients treated with chemotherapy (CT), several thousand times a year in our geographical area.

In order to take into account patient preferences and help clinical decision-making, this study will be conducted on the basis of self-administered questionnaires.

This research involves the administration/use of a product (PELGRAZ, Accord Healthcare) within its intended purpose. PELGRAZ prefilled syringe or prefilled pen are available on the European Union market.

The study will be carried out using a crossover design. Two modes of administration (syringe and pen) will be compared. Each subject will receive either the sequence syringe then pen, or pen then syringe.

The trial will be conducted among 150 cancer patients for whom a chemotherapy followed by the administration of pegfilgrastim is indicated.

The primary endpoint is a composite endpoint consisting of several parameters related to patient preference.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Patients with solid tumors, Hodgkin's lymphoma, non-Hodgkin's lymphoma and receiving myelosuppressive chemotherapy with a risk of NF of 10-20% (individual risk factors), or ≥ 20% (primary prevention of neutropenia) and receiving PELGRAZ ® in accordance with CPR
* Prediction of the risk of NF without filgrastim or pegfilgrastim determined according to the recommendations of the EORTC
* ECOG ≤ 2
* Free and informed consent obtained
* Patient affiliated to a social security system or beneficiary of such a scheme

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Patients receiving concurrent radiotherapy
* Second cancer treated with chemotherapy
* Participation in any other clinical trial within 30 days prior to recruitment
* Concomitant myelosuppressive therapy, e.g. ex. immunosuppressive therapy
* History of severe hypersensitivity reaction to drugs intended for use and/or drugs derived from E. coli

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients for whom a chemotherapy treatment followed by PELGRAZ administration is indicated
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
questionnaire | 120 days
  The primary endpoint is a composite endpoint consisting of several parameters related to patient preference

SECONDARY OUTCOMES:
questionnaire, specific questions | 120 days
  1. patient learning and empowerment during self-injection
  2. pain evaluation
  3. duration of treatment;
  4. patient satisfaction;
  5. overview of the health, physical and psychological conditions of the patient according to his own perception;

CONTACTS AND LOCATIONS:
Overall Officials: Alain TOLEDANO, MD, Principal Investigator — Institut Rafael
Locations (1):
- Institut Rafael, Levallois-Perret, Île-de-France Region, France

REFERENCES:
- [Derived] Scher N, Boudabous H, Partouche J, Rezaee-Vessal S, Ihout P, Rizzo C, Lamallem H, Bauduceau O, Darmon I, Bollet M, Draghi C, Toledano A. Enhancing patient-centered care: a randomized study on G-CSF administration preferences in chemotherapy-induced neutropenia. Support Care Cancer. 2024 Oct 22;32(11):743. doi: 10.1007/s00520-024-08929-x. PMID 39436413